CLINICAL TRIAL: NCT04378829
Title: Does the Platelet Count, Mean Platelet Volume and Platelet Distribution Width Change in COVID-19 Pandemic, ?
Brief Title: Platelet Count, Platelet, Mean Platelet Volume and Platelet Distribution Width in COVID-19
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Yasin Tire, Medical Doctor, Konya Meram State Hospital
Other Study IDs: COVID-19
Record Dates: First submitted 2020-05-03; First posted 2020-05-07 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Covid-19; Mean Platelet Volume; Platelet Destruction
MeSH Terms: conditions — COVID-19 | interventions — Platelet Count; Mean Platelet Volume

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ambulatory follow-up
  Interventions: Diagnostic Test: Platelet count, platelet, mean platelet volume and platelet distribution Width in COVID-19
- hospital follow-up
  Interventions: Diagnostic Test: Platelet count, platelet, mean platelet volume and platelet distribution Width in COVID-19
- intensive care unit follow-up
  Interventions: Diagnostic Test: Platelet count, platelet, mean platelet volume and platelet distribution Width in COVID-19

INTERVENTIONS:
Diagnostic Test: Platelet count, platelet, mean platelet volume and platelet distribution Width in COVID-19 — Platelet count, platelet, mean platelet volume and platelet distribution Width in COVID-19

SUMMARY:
The study will aim to investigate the relation of platelet count (PLT), mean platelet volume (MPV) and platelet distribution width (PDW) with other acute phase reactant c-reactive protein(CRP) in Coronavirus(COVID-19).

As a methodology, patients will be selected in records in one month from the online hospital system. Two groups will be divided before as need for mechanical ventilation or not. The latter comparison will be about three groups as an ambulatory follow-up, hospital follow-up, and intensive care unit follow-up. Parameters will be analyzed according to the groups.

DETAILED DESCRIPTION:
In this study, as a methodology, patients diagnosed with PCR test through the online system created for COVID-19 patients will be included in the study. These patients will be divided into 3 groups as outpatient follow-up, hospital follow-up and follow-up with a mechanical ventilator in intensive care. In addition, patients who have completed the 14-day treatment period, which is considered as the turning point time of the world health organization by looking at the patients 3 times, every 5-7 days, which is the accepted incubation period, will be included in the study. In these patients, hemoglobin, leukocyte, platelet, MPV, PDW and CRP values will be examined for 3 weekly measurements. Changes in COVID-19 disease follow-up and treatment of MPV and PDW values, which have not been studied so far, will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COVID-19, both PCR tests and computed tomography, as well as control hemogram and CRP tests at one week intervals will be included.

Exclusion Criteria:

* Those with suspicion of COVID-19, those who do not perform hemogram and c-reactive protein tests 3 times with one week intervals, those who do not have standard drug treatment will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study group will be selected from patients followed up in the 1-month period from the hospital online COVID-19 monitoring system.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2020-10-11 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Change in PDW and MPV parameters | 3 weeks totally tests.
  Expected increase or decrease in parameters according to the course of the disease

CONTACTS AND LOCATIONS:
Locations (1):
- Yasin Tire, Konya, Turkey (Türkiye)